CLINICAL TRIAL: NCT02025114
Title: A Phase IB/II, Open Label, Multicenter Study of Selumetinib Administered Orally in Combination With Gefitinib in Patients With EGFR-mutated Non-small Cell Lung Cancer Who Have Developed Acquired Resistance of EGFR Inhibitor Treatment
Brief Title: Selumetinib in Combination With Gefitinib in NSCLC Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201312070MIPC
Record Dates: First submitted 2013-12-24; First posted 2013-12-31 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: NSCLC, EGFR mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capsule (Experimental): The starting dose of selumetinib in combination with the standard dose of gefitinib (250mg QD) on a continuous dosing schedule will be 50mg QD. Total 3 doses of selumetinib will be tested (50mg QD, 50mg BID and 75mg BID).
  Interventions: Drug: selumetinib

INTERVENTIONS:
Drug: selumetinib — The starting dose of selumetinib in combination with the standard dose of gefitinib (250mg QD) on a continuous dosing schedule will be 50mg QD. Total 3 doses of selumetinib will be tested (50mg QD, 50mg BID and 75mg BID).

SUMMARY:
This is an open-label, non-randomized, multicenter phase Ib/II study, which is composed of a phase Ib dose escalation part and a phase II dose expansion part. Patients will receive selumetinib in combination with gefitinib 250mg daily. This study will enroll EGFR-mutated NSCLC patients who have developed acquired resistance to EGFR TKI treatment.

DETAILED DESCRIPTION:
he primary objective of the dose escalation part is to determine the MTD and/or RP2D of selumetinib in combination with gefinitib. Once MTD and/or RP2D has been determined in the phase Ib dose escalation phase, study drug selumetinib with combination of 250mg QD dose of gefitinib will be further evaluated in a phase II dose expansion phase of the study. The purpose of the dose expansion phase is to evaluate the efficacy of selumetinib in combination of gefitinib and to further characterize the safety, and tolerability of the combination.

20 patients will be required in the phase II period. In the expansion phase, 10 patients with T790M and 10 patients without T790M will be enrolled. It is assumed that 20% response rate is the target of clinical interest. If the true response rate is 20%, the probability of observing no responses in a random sample of 10 patients is 0.107. The false negative rate for detecting a true 20% response rate in each cohort is approximately 10%. Each cohort will be enrolled 10 patients to evaluate the efficacy; therefore 20 patients will be enrolled in dose expansion part. Patients treated at the MTD and/or RP2D during the phase Ib will be considered as part of the required number of patients in the phase II. Patients at the MTD or RP2D cannot contribute to the 20 patients require for phase II part.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any screening procedures.
2. ≥20 years of age.
3. Must have discontinued any previous anti-cancer and investigational therapy (excluding EGFR TKI) for at least 28 days or radiotherapy ≥14 days before study treatment administration, and must have recovered to Grade 1 from the adverse effects of such treatment before starting study treatment.
4. Life expectancy ≥3months.
5. ECOG performance status: 0-1.
6. Female patients of child-bearing potential should have a negative pregnancy test.
7. Required baseline laboratory status:

(1) Hemoglobin>9g/dL. (2) Platelet count≥100x109/L. (3) Absolute neutrophil count (ANC)≥1.5x109/L without growth factor support. (4) Total bilirubin 1.5x upper limit of normal (ULN). (5) AST/SGOT and/or ALT/SGPT 2.5x ULN. (6) Serum creatinine clearance >50 ml/min, by either Cockcroft-Gault formula or by 24-hour urine collection analysis.

8. Willing and able to comply with scheduled visits, treatment plan and laboratory tests.

9. In phase Ib part, lung cancer patients with disease progression after EGFR TKI and at least one line of chemotherapy. If less than 70 years of age, a platinum-based regimen must be included.

10. In phase II part, patients must be willing to perform a re-biopsy of the tumor at the time of study entrance and meet definition of acquired resistance criteria of Jackman's as follows:

(1) Previous treatment with EGFR TKI (gefitinib, erlotinib, afatinib, dacomitinib, AZD9291, or any EGFR TKI under investigation).

(2) Either or both of the followings:

1. A tumor harboring an EGFR mutation known to be associated with drug sensitivity (ie, exon 19 deletion , L858R, L861Q, G719X etc.).
2. Objectively clinical benefit from treatment with EGFR TKI as defined by either: Documented partial or complete response (RECIST or WHO) or Significant and durable(≥ 6months) clinical benefit (stable disease as defined by RECIST or WHO) after initiation of EGFR TKI.

   (3) Systemic progression of disease (RECIST or WHO) while on continuous treatment with EGFR TKI within the last 30 days.

   (4) No intervening systemic therapy between cessation of EGFR TKI and initiation the study treatment.

   Exclusion Criteria:
   1. Unable or unwilling to swallow capsules once or twice daily.
   2. Patients who had discontinued previous gefitinib treatment due to intolerance of side effects (such as diarrhea ≥CTCAE Grade 2, intolerable skin rash, ILD or AST/ALT elevation ≥ CTCAE Grade 3).
   3. Previous treatment of MEK, Ras, or Raf inhibitors or history of hypersensitivity to selumetinib, or any excipient agents.
   4. Symptomatic CNS metastases which are neurologically unstable or requiring increasing doses of steroids to control the CNS condition.
   5. Radiation therapy within 4 weeks prior to the first dose of study drug or limited field radiotherapy within 2 weeks prior to the start of study treatment. Any persistent side effect of prior radiotherapy must be resolved to Grade 1 prior to the first dose of study treatment.
   6. Any unresolved toxicity from previous anticancer therapy > Grade 1.
   7. Currently receiving any prohibited medications including vitamins supplements, and herbal supplements. Refer to Table 6.5 for a list of excluded medication.
   8. Unable to undergo an MRI or contrast CT procedures.
   9. Active HBV or HCV infection, HBV carrier can be enrolled if HBV DNA titer is low under antiviral treatment.
   10. Known history of HIV seropositivity. HIV testing is not required as part of this study.
   11. Undergone a bone marrow or solid organ transplant.
   12. Another malignancy diagnosed or treated within 5 years, except carcinoma in situ or skin cancer.
   13. Major surgery within 4 weeks prior to initiating study treatment, excluding the placement of vascular access.
   14. Cardiac conditions as follows:

   <!-- -->

   1. Uncontrolled hypertension (BP ≥150/95 mmHg despite medical therapy).
   2. Left ventricular ejection fraction <55% measured by echocardiography.
   3. Atrial fibrillation with a ventricular rate >100 bpm on ECG at rest.
   4. Symptomatic heart failure (NYHA grade II-IV), see Appendix A.
   5. Prior or current cardiomyopathy.
   6. Severe valvular heart disease.
   7. Uncontrolled angina (Canadian Cardiovascular Society grade II-IV despite medical therapy), see Appendix A.
   8. Acute coronary syndrome within 6 months prior to starting treatment". 15. Ophthalmological conditions as follows:

   <!-- -->

   1. Intra-ocular pressure >21 mmHg, or uncontrolled glaucoma (irrespective of intra-ocular pressure).
   2. Current or past history of central serous retinopathy or retinal vein occlusion.

   16. Past medical history of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis which required steroid treatment, pre-existing idiopathic pulmonary fibrosis or any evidence of clinically active interstitial lung disease.

   17. Pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (>5mIU/mL).

   18. Women of child-bearing potential, defined as all women physically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 30 more days after stopping study drug.

   19. Women are considered post-menopausal and not of child baring potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

   20. Sexually active males must use a condom during intercourse while taking the drug and for 30 more days after stopping study drug and should not father a child in this period. A condom is required to be used also by a vasectomized men in order to prevent delivery of the drug via seminal fluid.

   21. Any other condition that would, in the Investigator's judgment, contraindicate patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g. infection/inflammation, intestinal obstruction, unable to swallow medication, social/psychological issues, etc.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
To determine the MTD and/or RP2D | an expected average of 18 weeks
  Frequency and characteristics of DLTs to the selumetinib and gefitinib combination using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v.4.0. (an expected average of 18 weeks) If one patient experiences a DLT in a group of 3 or more evaluable patients, then the cohort will be expanded to include 6 evaluable patients. If only one DLT is observed in the complete cohort of 6 evaluable patients, then dose escalation may occur.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Patients will be followed up for 2 years(post disease progression)
  to estimate overall clinical activity of selumetinib combined with gefitinib in EGFR-mutated NSCLC patients who have acquired resistance to EGFR TKIs

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hsin Yang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (3):
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - Department of Oncology, National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei